CLINICAL TRIAL: NCT01920672
Title: Disrupted Sleep, Neuroendocrine Status and the Behavioral Symptoms of Alzheimer's Disease (AD)
Brief Title: Disrupted Sleep, Neuroendocrine Status and the Behavioral Symptoms of AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NA_00088139; P30NR014131 (NIH)
Record Dates: First submitted 2013-08-06; First posted 2013-08-12 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Timed Planned Activity (TPA) (Experimental): The TPA provides meaningful activities delivered at specific times in the daily diurnal cycle; it is theory-based, its components have been tested in pilot work; and it is portable and replicable (e..g, protocols are standardized). It involves involved 8 contacts (6 home visits and 2 phone calls) over 4 days. At baseline the CG completes the Pleasant Event Activity Survey. From the survey a careplan of meaningful activities are developed for the CG to administer. The suggested activities match the capabilities of an individual with moderate stage AD ie., based on repetitive motion (e.g., folding towels) and integrating multi-sensory stimulation (e.g., soft music, objects pleasant to touch). CG are instructed to introduce these activities during the late morning and early evening.
  Interventions: Behavioral: Timed Planned Activity
- Home Safety and Education Program (Active Comparator): The active comparator intervention will be delivered by interventionists who will provide social attention, empathy and engagement similar to that afforded to the experimental group. The length of time spent will be comparable to the length of time spent in the treatment arm. The attention-control group will involve 6 in-home visits in the afternoon and 2 brief telephone education sessions in the morning. Control group subjects will be provided a copy of Mace and Rabins, The 36-Hour Day, a well-known practical guidebook for families caring for AD patients. Each contact will provide helpful education based on a specific book chapter including information about home safety, health promotion, and advanced care planning
  Interventions: Behavioral: Home Safety and Education Program

INTERVENTIONS:
Behavioral: Timed Planned Activity
  Arms: Timed Planned Activity (TPA)
Behavioral: Home Safety and Education Program
  Arms: Home Safety and Education Program

SUMMARY:
Over 5 million Americans have Alzheimer's disease or a related dementia, a progressive and irreversible neurodegenerative condition, affecting also close to 15 million family caregivers (CG). Sleep efficiency in AD patients is severely impaired and complicated by frequent night awakenings and nocturnal restlessness. Untreated sleep disruption in AD patients is associated with increased rates of neuropsychiatric symptoms, daytime napping, 'sundowning' behaviors, cognitive and functional decline, and morbidity and mortality. The added strain of sleep disruption is the primary reason family caregivers make the decision to institutionalize AD patients. The circadian abnormalities in the sleep-wake cycle commonly observed in AD patients occur more often in individuals with hypothalamic/ pituitary/adrenal (HPA) axis hyperactivity. HPA axis hyperactivity may influence diurnal sleep-wake activity by diminishing an AD patient's ability to respond to external zeitgebers which, in turn, can further propagate HPA axis dysfunction. Thus, interventions to normalize diurnal HPA axis patterns may be beneficial in treating sleep-wake disturbances. Nonpharmacologic treatments are the first line therapy in AD patients with sleep wake problems, given the ineffective and potentially harmful effects of pharmacologic agents. Current clinical sleep hygiene practices in institutional (e.g., nursing home) settings holds promise for reducing disruptive sleep by reestablishing circadian patterns in HPA functioning. These interventions include use of timed and planned activities during daylight hours and creating a relaxing environment in the evening. However little systematic work has been done to determine the efficacy of these interventions in the home setting (where most individuals with AD reside).

We propose a pilot study to (a) characterize objective sleep parameters and behavioral symptoms of sleep-wake disturbance, and biological indicators of diurnal HPA axis activity in a sample of community residing older adults with AD: (b) examine the effects of timed and planned activities on subjective and objective characteristics of sleep, behavioral symptoms, and HPA status; and (c) evaluate measurement approaches in home-dwelling AD patients. Subjective (CG questionnaires) and objective (wrist actigraphy) characteristics of sleep and behavioral symptoms will be measured in fifty-four AD patients being cared for at home by a family. Patients and CG with then be randomized to receive an intervention of timed, planned activities (TPA) or attention control (AC) condition. We will also obtain diurnal measures of HPA activity including salivary cortisol and alpha amylase.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion/exclusion criteria are designed to obtain a sample of moderate stage AD patients because the sleep disruption we seek to assess occur most frequently at this stage. AD patients must: 1) have a diagnosis of probable AD (physician generated); 2) be over age 60; 3) be able to provide saliva samples; 4) be able to tolerate wrist actigraphy per caregiver report. Family caregivers must: 1) be English speaking; 2) have provided care for a minimum of 3 months; and 3) be the primary caregiver (self-identifies as providing the most day-to-day care).

Exclusion Criteria:

* To minimize the contribution of extraneous variables, subjects will be excluded for the following: regular use of medications with substantial known effects on the measurement of alpha amylase and cortisol (e.g. corticosteroids, interferons, beta-blockers, cytotoxic chemotherapy); major surgery in the past 3 months; history of major psychiatric and/or personality disorder; history of heavy cigarette smoking (e.g. >than 50 pack years); loss of a loved one in the past 3 months. Conditions known to affect measurement of sleep will also be excluded: use of sedatives/ hypnotics, Huntington's' disease, normal pressure hydrocephalus, Parkinson's disease, advanced heart failure (New York Heart Stage 3-4), morbid obesity (BMI > 35), and indications of restless legs syndrome or periodic limb movement disorder. We will exclude subjects screening positive for sleep apnea (actigraph/pulse oximetry oxygen desaturation index > 15).

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
total sleep time | 10 days
  total minutes of sleep

SECONDARY OUTCOMES:
Wake after sleep onset | 10 days
  number of episodes of wake activity after "lights out"

OTHER OUTCOMES:
Day/night sleep ratio | 10 days
  minutes of daytime sleep/ minutes of nighttime sleep

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Hodgson, PhD, Principal Investigator — Johns Hopkins Univeristy
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States